CLINICAL TRIAL: NCT03080714
Title: Topcon DRI OCT Triton Agreement and Precision Study
Brief Title: Triton Agreement and Precision Study
Status: Completed | Type: Observational
Sponsor: Topcon Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Organization: Topcon Corporation (Industry)
Other Study IDs: Triton AP
Record Dates: First submitted 2017-03-07; First posted 2017-03-15 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Healthy Eyes; Eye Diseases
Keywords: no known ocular pathology; Glaucoma; Retinal Disease
MeSH Terms: conditions — Eye Diseases; Glaucoma; Retinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Subjects Presenting With Normal Eyes: Subjects with no known ocular diseases will be scanned on the Topcon DRI OCT Triton (plus) device and 3D OCT-1 Maestro
  Interventions: Device: Topcon DRI OCT Triton (plus); Device: 3D OCT-1 Maestro
- Subjects presenting with Retinal Disease: Subjects with Retinal diseases will be scanned on the Topcon DRI OCT Triton (plus) device and 3D OCT-1 Maestro
  Interventions: Device: Topcon DRI OCT Triton (plus); Device: 3D OCT-1 Maestro
- Subjects presenting with Glaucoma: Subjects with Glaucoma will be scanned on the Topcon DRI OCT Triton (plus) device and 3D OCT-1 Maestro
  Interventions: Device: Topcon DRI OCT Triton (plus); Device: 3D OCT-1 Maestro

INTERVENTIONS:
Device: Topcon DRI OCT Triton (plus) — The Topcon DRI OCT Triton (plus) is an OCT machine used for diagnostic purposes
Device: 3D OCT-1 Maestro — The 3D OCT-1 Maestro is an OCT machine used for diagnostic purposes

SUMMARY:
To Compare the agreement and precision between the Topcon DRI OCT Triton and the 3D OCT-1 Maestro with RDB.

DETAILED DESCRIPTION:
The objectives of this study are to compare the agreement and precision between Topcon DRI OCT Triton and 3D OCT-1 Maestro with RDB by measuring the thickness layers.

ELIGIBILITY:
Inclusion Criteria for Normal Group

1. Subjects 18 years of age or older on the date of informed consent
2. Subjects able to understand the written informed consent and willing to participate as evidenced by signing the informed consent
3. Subjects presenting at the site with normal eyes bilaterally (cataracts are acceptable)
4. IOP ≤ 21 mmHg bilaterally
5. BCVA 20/40 or better bilaterally

Exclusion Criteria for Normal Group

1. Subjects unable to tolerate ophthalmic imaging
2. Subjects with ocular media not sufficiently clear to obtain acceptable OCT images
3. HFA visual field (24-2 Sita Standard, white on white) result unreliable (based on manufacturer's recommendation), defined as fixation losses > 20% or false positives > 33%, or false negatives > 33%
4. Visual field defects consistent with glaucomatous optic nerve damage based on at least one of the following two findings:

   1. On pattern deviation (PD), there exists a cluster of 3 or more points in an expected location of the visual field depressed below the 5% level, at least 1 of which is depressed below the 1% level;
   2. Glaucoma hemi-field test "outside normal limits."
5. Narrow angle
6. History of leukemia, dementia or multiple sclerosis
7. Concomitant use of hydroxychloroquine and chloroquine

Inclusion Criteria for Glaucoma Group

1. Subjects 18 years of age or older on the date of informed consent
2. Subjects able to understand the written informed consent and willing to participate as evidenced by signing the informed consent
3. BCVA 20/40 or better in the study eye
4. Visual field defects consistent with glaucomatous optic nerve damage based on at least one of the following two findings:

   1. On pattern deviation (PD), there exists a cluster of 3 or more points in an expected location of the visual field depressed below the 5% level, at least 1 of which is depressed below the 1% level;
   2. Glaucoma hemi-field test "outside normal limits."
5. Glaucomatous optic nerve damage as evidenced by any of the following optic disc or retinal nerve fiber layer structural abnormalities:

   1. Diffuse thinning, focal narrowing, or notching of the optic disc rim, especially at the inferior or superior poles with or without disc hemorrhage;
   2. Localized abnormalities of the peripapillary retinal nerve fiber layer, especially at the inferior or superior poles; or
   3. Optic disc neural rim asymmetry of the two eyes consistent with loss of neural tissue

Exclusion Criteria for Glaucoma Group

1. Subjects unable to tolerate ophthalmic imaging
2. Subject with ocular media not sufficiently clear to obtain acceptable OCT images
3. HFA visual field (24-2 Sita Standard, white on white) result unreliable, defined as fixation losses > 20% or false positives > 33%, or false negatives > 33% in the study eye
4. Presence of any ocular pathology except glaucoma in the study eye (cataracts are acceptable)
5. History of leukemia, dementia or multiple sclerosis
6. Concomitant use of hydroxychloroquine and chloroquine

Inclusion Criteria for Retina Disease Group

1. Subjects 18 years of age or older on the date of informed consent
2. Subjects able to understand the written informed consent and willing to participate as evidenced by signing the informed consent
3. Subjects presenting at the site with retinal disease
4. IOP ≤ 21 mmHg in the study eye
5. BCVA 20/400 or better in the study eye
6. Diagnosis of some type of retinal pathology by investigator, may include, but not limited to: Macular Degeneration, Diabetic Macular Edema, Diabetic Retinopathy, Macular Hole, Epiretinal Membrane, Cystoid Macula Edema, and others

Exclusion Criteria for Retinal Disease Group

1. Subjects unable to tolerate ophthalmic imaging
2. Subject with ocular media not sufficiently clear to obtain acceptable OCT images
3. Presence of glaucoma or any ocular pathology other than a Retinal pathology (e.g., cornea pathology) in the study eye (cataracts are acceptable)
4. Narrow angle in the study eye
5. History of leukemia, dementia or multiple sclerosis
6. Concomitant use of hydroxychloroquine and chloroquine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects presenting with Glaucoma, Retinal Diseases, or with no Ocular Pathology.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Retinal Thickness | 1 Minute
  The thickness of the macula layer

CONTACTS AND LOCATIONS:
Overall Officials: Charles Riesman, MS, Study Chair — Topcon Corporation
Locations (1):
- Fischer Laser Eye Center, Willmar, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No